CLINICAL TRIAL: NCT02359032
Title: A Phase 1 Combined Single and Multiple Ascending Oral Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASP6858 in Healthy Subjects
Brief Title: A Combined Single and Multiple Ascending Dose Study of ASP6858 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 6858-CL-0001; 2014-003735-18 (EudraCT Number)
Record Dates: First submitted 2015-02-04; First posted 2015-02-09 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteers
Keywords: Healthy subjects; Pharmacokinetics of ASP6858; ASP6858; Pharmacodynamics of ASP6858

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1: ASP6858 single ascending dose (Experimental): ASP6858 arm
  Interventions: Drug: ASP6858
- Part 1: Placebo single ascending dose (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo
- Part 1: ASP6858 single ascending dose (fasting cohort) (Experimental): ASP6858 arm
  Interventions: Drug: ASP6858
- Part 2, Sequence 1: ASP6858 multiple ascending dose & placebo (Experimental): ASP6858 and placebo arm
  Interventions: Drug: ASP6858; Drug: Placebo
- Part 2, Sequence 2: ASP6858 multiple ascending dose & placebo (Experimental): ASP6858 and placebo arm
  Interventions: Drug: ASP6858; Drug: Placebo

INTERVENTIONS:
Drug: ASP6858 — Oral tablets
  Arms: Part 1: ASP6858 single ascending dose; Part 1: ASP6858 single ascending dose (fasting cohort); Part 2, Sequence 1: ASP6858 multiple ascending dose & placebo; Part 2, Sequence 2: ASP6858 multiple ascending dose & placebo
Drug: Placebo — Oral tablets
  Arms: Part 1: Placebo single ascending dose; Part 2, Sequence 1: ASP6858 multiple ascending dose & placebo; Part 2, Sequence 2: ASP6858 multiple ascending dose & placebo

SUMMARY:
The purpose of this study is evaluate the safety and tolerability of single and multiple ascending oral doses of ASP6858. This study will also evaluate the pharmacokinetics (PK) of ASP6858 and its metabolites as well as the effect of food to the PK of ASP6858. The study will also evaluate the pharmacodynamics of ASP6858.

DETAILED DESCRIPTION:
This study has 2 parts: Part 1 is a placebo-controlled, single ascending dose study where male only subjects will be residential for 5-8 days (Part 1 will also include an open-label, food effect section); and Part 2 is a placebo-controlled, randomized, 2-way crossover, multiple ascending dose study where male and female subjects will be residential for 14-17 days for each treatment period. There will be a washout period between the 2 periods in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Healthy male subject, 18 to 55 years of age, inclusive, at screening. Part 2: Healthy male or female subject, 18 to 55 years of age, inclusive, at screening.
* Subject has a body mass index range of 18.5 to 30.0 kg/m2, inclusive, and weighs at least 50 kg, at screening.
* Subject has stable eating habits and weight (± 2 kg) over the last 4 weeks prior to screening.
* Subject is willing to comply strictly with the diet applied during the clinical study.
* Subject agrees not to participate in another interventional study while participating in the present clinical study, defined as signing the informed consent form until completion of the last study visit.

Exclusion Criteria:

* Subject had prior upper gastric, gastroduodenal, pancreatic or small intestinal surgery.
* Subject has lactose intolerance, gluten sensitivity or other condition with significant nutritional malabsorption.
* Female subject who has been pregnant within 6 months prior to screening assessment or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to ASP6858 or any components of the formulations used.
* Subject has any of the liver chemistry tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase, gamma glutamyl transferase, total bilirubin [TBL]) above the upper limit of normal (ULN). In such a case the assessment may be repeated once on day -1 (in part 2: treatment period 1 only).
* Subject has any clinically significant history of allergic conditions.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to admission to the clinical unit (in part 2: treatment period 1 only).
* Subject has any clinically significant abnormality following the investigator's review of the physical examination, ECG and protocol-defined clinical laboratory tests at screening or admission to the clinical unit (in part 2: treatment period 1 only).
* Subject has a mean pulse < 40 or > 90 bpm; mean systolic blood pressure > 140 mmHg; mean diastolic blood pressure > 90 mmHg (vital signs measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically) at screening and day -1 (in part 2: treatment period 1 only). If the blood pressure exceeds the limits above, 1 additional triplicate can be taken.
* Subject has a mean corrected QT interval using Fridericia's formula > 430 ms (for male subjects) and > 450 ms (for female subjects) on day -1 (in part 2: treatment period 1 only). If these limits are exceeded, 1 additional triplicate ECG can be taken.
* Subject uses any prescribed or nonprescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to study drug administration, except for occasional use of paracetamol (up to 2 g/day) and except for use of contraceptives or hormone replacement therapy.
* Subject has a history of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the clinical unit (in part 2: first admission).
* Subject has a history of drinking more than 21 units (male subjects) or 14 units (female subjects) of alcohol per week (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months prior to admission to the clinical unit (in part 2: first admission).
* Subject uses any drugs of abuse within 3 months prior to admission to the clinical unit (in part 2: first admission).
* Subject uses any inducer of metabolism (e.g., barbiturates, rifampin) in 1 month prior to admission to the clinical unit (in part 2: first admission).
* Subject had significant blood loss, donated 1 unit (500 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to admission to the clinical unit (in part 2: first admission).
* Subject has a positive serology test for hepatitis B surface antigen, hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies or antibodies to human immunodeficiency virus type 1 (HIV-1) and/or type 2 (HIV-2) at screening.
* Subject participated in any clinical study or has been treated with any investigational drugs within 3 months or 5 terminal half-lives, whichever is longer, prior to screening.
* Subject is unable to communicate, read and understand English, or has any other condition which, in the investigator's opinion, makes the subject unsuitable for clinical study participation.
* Subject is an employee of the Astellas Group, a Clinical Research Organization or other vendor involved in the clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by adverse events | Part 1 = up to 17 days; Part 2 = up to 50 days
Safety as assessed by vital signs | Part 1 = up to 17 days; Part 2 = up to 50 days
  blood pressure, pulse rate, body temperature
Safety as assessed by clinical laboratory tests | Part 1 = up to 17 days; Part 2 = up to 50 days
  Biochemistry, hematology, urinalysis
Safety as assessed by 12-lead electrocardiogram (ECG) | Part 1 = up to 17 days; Part 2 = up to 50 days
Safety as assessed by continuous cardiac monitoring | Part 1 = Days 1-4; Part 2 = Day 10
  Part 1 = N/A for fasting cohort
Safety as assessed by coagulation parameters: aPTT, PT | Part 1 = up to 17 days; Part 2 = up to 50 days
  Activated partial thromboplastin time (aPTT); Prothrombin time (PT)
Safety as assessed by body weight (Part 2) | up to 50 days

SECONDARY OUTCOMES:
Secondary Outcome Title: Pharmacokinetic profile of ASP6858 (plasma): AUCinf, AUC5, AUC14, AUC24, AUClast, tlag, tmax, Cmax, t½, Vz/F, CL/F (Part 1) | Day 1
  Cumulative amount of study drug excreted into urine from time of dosing extrapolated to time infinity (AUCinf); Area under the concentration-time curve from the time of dosing to 5 hours postdose (AUC5); Area under the concentration-time curve from the time of dosing to 14 hours postdose (AUC14); Area under the concentration-time curve from the time of dosing to 24 hours postdose (AUC24); Area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast); Time prior to the time corresponding to the first measurable (nonzero) concentration (tlag); Time of maximum concentration (tmax); Maximum concentration (Cmax); Terminal elimination half-life (t1/2); Apparent volume of distribution during the terminal elimination phase after single or multiple extravascular dosing (Vz/F); Apparent total systemic clearance after single or multiple extravascular dosing (CL/F)
Pharmacokinetic profile of ASP6858 metabolite M1 and M2 (plasma): AUCinf, AUC5, AUC14, AUC24, AUClast, tlag, tmax, Cmax, t½, MPR (Part 1) | Day 1
  Metabolite to parent ratio (MPR)
Pharmacokinetic profile of ASP6858, metabolites M1 and M2 (urine): Ae24, Ae24%, Aelast, Aelast%, Aeinf, Aeinf%, CLR (Part 1) | Day 1
  Percentage of study drug excreted into urine from time of dosing to 24 hours postdose (Ae24%); Cumulative amount of study drug excreted into urine from time of dosing up to the collection time of the last measurable concentration (Aelast); Percentage of study drug dose excreted into urine from time of dosing up to the collection time of the last measurable concentration (Aelast%); Cumulative amount of study drug excreted into urine from time of dosing extrapolated to time infinity (Aeinf); Renal clearance (CLR)
Pharmacokinetic profile of ASP6858 and metabolites M1 and M2 (plasma): Ctrough, morning (Part 2) | Days 3, 6 and 9
  Concentration immediately prior to morning dosing (Ctrough, morning)
Pharmacokinetic profile of ASP6858 and metabolites M1 and M2 (plasma): tmax, Cmax, AUC5, PTR, AUC14, t1/2, AUC24 (Part 2) | Day 10
  Peak trough ratio (PTR)
Pharmacokinetic profile of ASP6858 (plasma):Vz/F, CL/F | Day 10
Pharmacokinetic profile of ASP6858 metabolites M1 and M2 (plasma): MPR, MPR24 | Day 10
  Metabolite to parent ratio from the time of dosing to 24 hours postdose (MPR24)
Pharmacokinetic profile of ASP6858 and metabolites M1 and M2 (urine): Ae24, Ae24%, CLR,24 | Day 10
Pharmacodynamic profile (urine): 24UUN and UNA | Day 8-10
  24-hour urinary urea nitrogen (24UUN); urinary nitrogen appearance (UNA)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Site GB44001, Harrow, United Kingdom